CLINICAL TRIAL: NCT02033785
Title: Prospective Cohort Study of Holmium Laser Prostatectomy For Observing Functional Changes in Benign Prostate Hyperplasia Patients
Brief Title: Functional Changes of Urogenital System After Holmium Laser Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Seung-Ju Lee, Senior researcher, The Catholic University of Korea
Other Study IDs: L201401N1; VC13OISI0222 (Other: IRB of St. Vincent's Hospital)
Record Dates: First submitted 2014-01-07; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Prostatic Hyperplasia
Keywords: Prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Holmium laser prostatectomy will enhance voiding function.

Holmium laser prostatectomy will enhance sleep quality.

Holmium laser prostatectomy will enhance renal function.

Holmium laser prostatectomy will enhance erectile function.

Holmium laser prostatectomy will enhance the health-related quality of life.

DETAILED DESCRIPTION:
Check urodynamic parameters for voiding function evaluation Check low urinary tract symptoms (IPSS: international prostate symptom score) for voiding function evaluation Check Pittsburgh Sleep Quality Index for sleep quality evaluation Check estimated glomerular filtration rate and urine protein/creatinine ratio for renal function evaluation Check International Index of Erectile Function score (IIEF-5) for erectile function evaluation Check nocturnal penile tumescence parameters for erectile function evaluation Check 36-Item Short- Form Health Survey (SF-36) for evaluation of the health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Prostate size over 30 cc by transrectal ultrasonography
* prostate-specific antigen level less than 10 ng/ml
* International prostate symptom score more than 7
* At least one of followings: Bladder outlet obstruction index > 40, maximal flow rate < 10 cc/sec, postvoid residual urine >100cc or schäfer grade II or more

Exclusion Criteria:

* Patients who do not want surgery
* Evidence of prostate cancer or bladder cancer during evaluation or treatment
* All of followings: Bladder outlet obstruction index is less than 40, maximal flow rate is 10 or more cc/sec, postvoid residual urine is less than 100cc and schäfer grade II or less
* Major depressive disorder, Dementia, Parkinson's disease, Neurological deficits
* History of pelvic radiation therapy
* Poorly controlled diabetes mellitus or hypertension

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Maximal flow rate | 3 months
  This parameter can be obtained from urodynamic study.
Maximal detrusor pressure | 3 months
  This parameter can be obtained from urodynamic study.
Bladder outlet obstruction index | 3 months
  This parameter can be obtained from urodynamic study.
schäfer grade | 3 months
  This parameter can be obtained from urodynamic study.
Compliance | 3 months
  This parameter can be obtained from urodynamic study.

SECONDARY OUTCOMES:
Maximal flow rate | 12 months
  This parameter can be obtained from urodynamic study.
Maximal detrusor pressure | 12 months
  This parameter can be obtained from urodynamic study.
Bladder outlet obstruction index | 12 months
  This parameter can be obtained from urodynamic study.
schäfer grade | 12 months
  This parameter can be obtained from urodynamic study.
Compliance | 12 months
  This parameter can be obtained from urodynamic study.

OTHER OUTCOMES:
international index of erectile function | 3 months
international index of erectile function | 12 months
normalized rigidity activity unit in penile tip | 3 months
  This parameter can be obtained from nocturnal penile tumescence test.
normalized rigidity activity unit in penile tip | 12 months
  This parameter can be obtained from nocturnal penile tumescence test.
normalized rigidity activity unit in penile base | 3 months
  This parameter can be obtained from nocturnal penile tumescence test.
Estimated glomerular filtration rate | 3 months
Estimated glomerular filtration rate | 12 months
Urinary protein to creatinine ratio | 3 months
Urinary protein to creatinine ratio | 12 months
International prostate symptom score | 3 months
International prostate symptom score | 12 months
Pittsburgh Sleep Quality Index | 3 months
Pittsburgh Sleep Quality Index | 12 months
Health-related quality of life, short form 36 score | 3 months
Health-related quality of life, short form 36 score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Ju Lee, Study Chair — The Catholic University of Korea; Dong Sup Lee, Principal Investigator — The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, The Catholic University of Korea, Suwon, Gyeonggi-do, South Korea